CLINICAL TRIAL: NCT00159341
Title: Cigarette Smoke Nasal and Whole Blood Challenge in Patients With COPD
Brief Title: Cigarette Smoke Nasal and Whole Blood Challenge in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Dr Trevor Hansel, NHLI Clinical Studies Unit
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 05/Q0404/84
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Lung Diseases, Obstructive
Keywords: cigarette smoke; nasal; whole blood; cytokines; chemokines; nasal fluid; filter paper
MeSH Terms: conditions — Lung Diseases, Obstructive; Cigarette Smoking | interventions — Nasal Lavage; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Nasal lavage — Nasal lavage was carried out at specified timepoints
Procedure: Nasal filter paper — Nasal filter paper was placed at specified timepoints
Procedure: Blood sampling — Blood sampling was performed as a routine safety check

SUMMARY:
This is a clinical research study to assess whether after exhaling a single cigarette smoke through the nose there are changes in the inflammatory cells and proteins of nasal secretions.

A single blood sample from each subject will be stimulated with cigarette smoke in the laboratory to see the effects on inflammatory blood cells.

Comparison of findings between smokers with COPD and "Healthy" smokers will be carried out.

We hypothesize that some subjects have amplified inflammatory response to a single cigarette, and these will be those subjects who develop chronic obstructive pulmonary disease (COPD) after decades of smoking. We hope to develop an acute challenge model that relates to the causation of COPD. When studying the effects of new drugs, these may be detected in small numbers of patients in a challenge situation, when we would need to study many more unchallenged patients to demonstrate drug effects. In clinical research on asthma and allergy, the nasal allergen challenge has been a very successful model, and we hope to validate a comparable model for COPD.

DETAILED DESCRIPTION:
Introduction Chronic obstructive pulmonary disease (COPD) is a common respiratory disease that causes widespread morbidity and mortality, the Global Burden of Disease Study estimating COPD to be currently the sixth most common cause of death worldwide. Decades of cigarette smoking is by far the major contributing factor, and this causes a range of respiratory disorders; including chronic bronchitis, obstructive bronchiolitis, emphysema, and pulmonary vascular disease. Medical treatment of COPD is largely palliative; involving smoking cessation, use of inhaled bronchodilators, and long term oxygen therapy for respiratory failure. Recently, it has been recognised that those smokers who develop COPD have amplification of inflammation compared with "healthy smokers", and that there is the urgent need to develop new challenge models to assess why COPD develops in some heavy smokers.

Cigarette Smoke Nasal Challenge Model The nose is an accessible part of the respiratory system, from which it is possible to obtain tissue exudates and cell brushings in a non-invasive manner. A comprehensive review of the extensive clinical research experience with these nasal methodologies has recently been published. There is also the insight that patients with COPD commonly have inflammation of both the airways and nasal passages, with a similar type of inflammatory infiltrate in lower and upper airways. In COPD the inflammation is predominantly involving neutrophils and macrophages, as opposed to the increase in mast cells and eosinophils characteristic of asthma.

It has long been recognised that there is a strong functional and immunological relationship between the nose and bronchi, especially in terms of infiltrating leukocytes and inflammatory mediators when comparing allergic rhinitis and allergic asthma. The upper and lower airways have related respiratory epithelium and similar responses to allergen challenge.

The nasal and bronchial mucosa of smokers with COPD have been demonstrated to be infiltrated with CD8+ T lymphocytes and neutrophils. This corresponds to the presence of nasal symptoms during exacerbations of COPD, and sputum and nasal levels of IL-8 are correlated in COPD.

In order to sample nasal exudates for allergic inflammatory mediators, the classical methods of nasal lavage are those described by Naclerio et al., the nasal pool method of Greiff et al., and the use of a Foley's catheter by Grünberg and colleagues. Lavage is performed with saline at volumes of between 1 and 10ml. The repeatability and validity of different nasal lavage methods have been compared.

Tommy Sim and colleagues have developed the use of filter paper strips, that are placed on the turbinates to absorb nasal secretions. The nasal filter paper method has the advantage of directly sampling nasal secretions which are less diluted and can therefore pick up protein signals which are below the detection limits of nasal lavage. The matrix or filter paper method has been used to measure chemokines and cytokines after NAC.

Cells samples may be obtained from the nasal mucosal using small nylon dental flossing brushes which are gently rotated over the epithelium, and then the attached cells are dislodged in balanced salt solution. It has been demonstrated that nasal brushing can be used as an alternative to nasal biopsy [24], whilst nasal brush supernatants can be analysed for cytokine release [25]. An alternative method is to employ nasal mucosal scrapings using a plastic curette (Rhinoprobe, Arlington Scientific, Utah). Nasal brushing and scraping causes some discomfort but does not require local anaesthesia. Nasal biopsy is generally performed from the lower edge of the inferior turbinate by a specialist. This is a traumatic procedure that requires careful local anaesthesia, but a specimen of mucosal epithelium with basement membrane and submucosal tissue is obtained.

Nasal allergen challenge (NAC) is of proven benefit to test novel anti-inflammatory therapy for allergic rhinitis and asthma.

NAC has advantages over inhaled allergen challenge since it is easier to recruit subjects, it is less invasive, and repeated tissue samples are readily obtained. Small numbers of patients can be given even single doses of therapy, and the anti-inflammatory and clinical effects on NAC responses noted. Using these challenge methods in phase II of drug development for asthma and allergic rhinitis it is possible to provide an early and reliable "Go/No Go" decision before embarking on large-scale, long-term and costly phase III studies.

We hope to develop an analogous challenge model for COPD by assessing effects of nasal challenge with cigarette smoke.

A major challenge is to develop phase IIa clinical pharmacology designs that can be used to assess anti-inflammatory drugs being developed for COPD. Nasal epithelial and inflammatory responses to ozone exposure have been much studied [31-39]. Indeed COPD is characterised by chronic inflammation with an imbalance in oxidant/antioxidant levels, and systemic inflammation may trigger local exercise-induced oxidative stress.

Three year clinical trials involving thousands of patients have found that inhaled corticosteroids do not affect the accelerated rate loss of lung function in COPD. Furthermore, ongoing phase III trials with oral phosphodiesterase type 4 (PDE4)inhibitors are also unconvincing, despite the initial smaller studies looking promising. There is clearly the compelling need to develop non-invasive biomarkers and clinical challenge models for use in phase II clinical pharmacology studies to enable reliable assessment of the effects of anti-inflammatory therapy in COPD.

Use of nasal challenge models coupled to sensitive biomarkers and clinical endpoints could perhaps be used to establish clinical efficacy of new drugs for COPD in small scale studies. Novel therapies have the potential to selectively inhibit various cell types and particular mediators involved in diverse inflammatory diseases. We believe that nasal allergen challenge has advantages over inhaled challenge: safety, repeat non-invasive sampling.

In the future this will ensure that nasal challenge will play a growing role in clinical pharmacology assessment of anti-inflammatory therapy. Major efforts are ongoing to develop nasal challenge models to mimic the inflammation found in COPD, that can be used in clinical pharmacology assessment of new anti-inflammatory drugs.

Whole Blood Challenge in vitro with Cigarette Smoke We shall stimulate blood samples in the laboratory in an in vitro manner with a cigarette smoke extract. The cigarette smoke extract is produced in a fume cabinet ensuring the safety of laboratory personnel. Cigarette smoke contains many toxic compounds including free radicals and oxidants. Cigarette smoke conditioned medium (CSCM) is made by bubbling the smoke from burning cigarettes through buffered salt solution, and this can be used to stimulate cells in vitro. Cigarette smoke extract has been shown to be cytotoxic to an alveolar type II cell-derived line and this effect can be blocked by N-acetyl cysteine a scavenger of oxidants. {Hoshino, Mio, et al. 2001 7463 /id}. We have developed methods of assessing neutrophil CD11b upregulation in response to stimulation with cytokines and chemokines. CD11b is a cell surface receptor on leukocytes that is mobilised from intracellular stores when cells are stimulated. Surface CD11b can be measured using fluorescent labelled antibodies and flow cytometry. We have developed a method of stimulating whole blood with CSCM which produces a 200% increase in CD11b upregulation after incubation for 20 minutes. This effect is further increased if plasma is removed from the whole blood prior to stimulation, and the effect can be partially inhibited by the presence of reduced glutathione. COPD patients and smokers have been shown to have decreased antioxidant capacity in their plasma. We aim to compare neutrophil responses to CSCM stimulation in whole blood, and washed blood where the plasma has been removed, to compare neutrophil responsiveness between COPD patients and smokers and possible anti-oxidant effects of plasma.

Overview of planned research

Two characterised matched groups of smokers with COPD and "healthy" smokers that do not have lung disease will be enrolled for this study. Each group will comprise 8 subjects. Each subject will be required to make 2 visits to the NHLI Clinical Studies Unit as follows:

Visit 1 : Screening During screening, candidates for the study will be fully informed about the nature of the study and possible AEs. Candidates must read the consent form and sign the document after the investigator has answered all questions to the candidate's satisfaction. Further procedures can begin only after the consent form has been signed. Two original informed consent form copies will be signed by the subject. An original signed consent form will be retained by the investigator and the second original will be given to the candidate to take home.

Candidates will be evaluated for entry into the study according to the stated inclusion and exclusion criteria. The following procedures will be performed to establish each candidate's general health and qualifications for enrollment into the study:

* Obtain signed, written informed consent
* Record medication history over the past 30 days Record medical history, including smoking status
* Perform a physical examination of heart, lung and nose
* Pregnancy test for female subjects of child bearing age
* Conduct spirometry and test reversibility
* Review inclusion and exclusion criteria

The investigator will evaluate the results of all examinations including clinical laboratory tests and will determine each candidate's suitability for the study. When the subject is suitable for the study, a blood sample (10mls) will be taken for cigarette smoke whole blood challenge.

Visit 2: Nasal smoke challenge Each subject will be allowed to smoke at least 5 cigarettes between 9am to 9pm the day before attending the unit, and on the previous 7 days. On the study day, each patient will be asked to smoke a single cigarette but exhaling through the nose.

Following this cigarette challenge, we will carry out the following procedures over a period of 8 hours (pre(x2), 1h, 2h, 3h, 4h,6h and 8h):

1. Nasal lavage consists of washing the nose of 5ml (a teaspoon) of warm salt solution. This solution is gently passed from a syringe through a hollow "olive" into the end of the left nostril. The fluid does not enter the sinuses nor pass down the back of the nose. A total of 2 flushes will be carried out at each timepoints.
2. Nasal filter paper consists of a 7mm x 30mm strips of paper that are gently place inside the end of the right nostril. They are left there for up to2 minutes until they are moist with nasal secretions.
3. A cannula will be inserted to enable blood to be taken at the above time points for serum analysis of cytokines and chemokines.
4. Pregnancy test for female subjects of child bearing age only.

As part of the study, subjects will be informed of the harmful effects of cigarette smoking, and advised of the need to stop smoking. Subjects will be offered smoking classes to help them stop smoking. It is anticipated that the study day will be set as the quit date for subjects.

ELIGIBILITY:
Inclusion Criteria (COPD Smokers):

* Smokers currently on at least 5 cigarettes per day, with a history of >10 pack years
* Post-bronchodilator FEV1 >30% of predicted and < 80% of predicted
* Pre-bronchodilator FEV1/FVC of <70%
* With or without chronic simple bronchitis

Exclusion criteria (COPD Smokers):

* History of asthma, allergy (including rhinitis/eczema)
* Reversibility : an increase in FEV1 that is >400ml from the baseline pre- bronchodilator value (bronchodilate with salbutamol 400g delivered from a metered dose inhaler (MDI) into a spacer).

Inclusion criteria (for "Healthy" Smokers):

* Smokers currently on at least 5 cigarettes per day, with a history of >10 pack years
* FEV1 >90% of predicted, FEV1/FVC of >70%
* Cannot have chronic simple bronchitis
* Age, sex, smoking history matched to COPD Smokers

Exclusion criteria (for "Healthy" Smokers):

* History of asthma, allergy (including rhinitis/eczema
* Reversibility: an increase in FEV1 that is both >400ml from the baseline pre-bronchodilator value (bronchodilate with salbutamol 400mcg delivered from a metered dose inhaler (MDI) into a spacer)P
* Pregnancy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2005-09; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Changes in the cytology and inflammatory mediator content of nasal exudates | Single timepoint

SECONDARY OUTCOMES:
Comparison of nasal inflammatory response to smoke in patients with COPD with relevant controls | Single timepoint
Comparison of inflammatory response in blood following cigarette smoking in patients with COPD and relevant controls | Single timepoint
Comparison of nasal challenge with blood challenge | Single timepoint
Develop a nasal challenge model to test novel anti-inflammatoy therapies for COPD | Single timepoint
Identification of potential biomarkers for therapeutic trials in COPD | Single timepoint
Definition of novel drug targets for potential new anti-inflammatory therapies | Single timepoint

CONTACTS AND LOCATIONS:
Overall Officials: Trevor T Hansel, BSc MSc PhD, Principal Investigator — National Heart & Lung Institute, Imperial College London
Locations (1):
- National Heart & Lung Institue Clinical Studies Unit, Imperial College London, London, United Kingdom

REFERENCES:
- [Result] - Vachier I et al.Inflammatory features of nasal mucosa in smokers with and without COPD. Thorax 2004; 59:303-307. - Naclerio RM et al. Mediator release after nasal airway challenge with allergen. Am Rev Respir Dis 1983; 128:597-602. - Greiff L et al. The 'nasal pool' device applies controlled concentrations of solutes on human nasal airway mucosa and samples its surface exudations/secretions. Clin Exp Allergy 1990; 20:253-259. - Alam R et al. Development of a new technique for recovery of cytokines from inflammatory sites in situ. J Immunol Methods 1992; 155:25-29. - Weido AJ et al. Intranasal fluticasone propionate inhibits recovery of chemokines and other cytokines in nasal secretions in allergen-induced rhinitis. Ann Allergy Asthma Immunol 1996; 77:407-415. - Meltzer EO, Jalowayski AA. Nasal cytology in clinical practice. Am J Rhinol 1988; 2:47-54. - Fishwick D et al. Immunologic response to inhaled endotoxin: changes in peripheral cell surface markers in normal individuals. J Occup Environ Med 2004; 46:467-472. - Mudway IS, Kelly FJ. An investigation of inhaled ozone dose and the magnitude of airway inflammation in healthy adults. Am J Respir Crit Care Med 2004; 169:1089-1095. - Rahman I et al. Glutathione, stress responses, and redox signalling in lung inflammation. Antioxidants & Redox Signalling 2005; 7:42-59. - Koechlin C et al. Does systemic inflammation trigger local exercise-induced oxidative stress in COPD? Eur Respir J 2004; 23:538-544.
- See also: Imperial College London website — http://www.ic.ac.uk